CLINICAL TRIAL: NCT00715754
Title: Antecedents of Obesity: Fetal Measures of Adiposity, "A Plan for Obesity Disaster Management"
Brief Title: Antecedents of Obesity: Fetal Measures of Adiposity
Acronym: FEMA
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 18858
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to study whether fetal biometrics obtained by 2-D ultrasound can predict infant adiposity by air displacement plethysmography at birth.

ELIGIBILITY:
Inclusion Criteria:

* Infants of mothers between the ages of 18 and 45, planning child birth at the University of Utah Hospital, and willing to provide parental permission for the child to participate in the study.

Exclusion Criteria:

* Infants of mothers under the age of 18, over the age of 45, planning child birth at another facility other than the University of Utah Hospital, or who are not willing to provide permission for the child to participate in the study.

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born at the University of Utah Hospital, whose mothers received prenatal care also at the University of Utah Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Moyer-Mileur, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Infants: One group comprised all infants evaluated.
Period: Overall Study
Arm/Group | All Infants
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infants
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Infant Adiposity at 24-72 Hours Following Birth
Description: Adiposity as measured by air displacement plethysmography
Time Frame: 24-72 hours following birth
Measure: Mean (Full Range); unit: Percentage of total body weight
Groups:
- Newborn Infants: Newborn Infants
Arm/Group | Newborn Infants
Number analyzed (Participants) | 47
Percentage of total body weight | 11 [3 to 21]

2. Primary Outcome: Fetal Abdominal Circumference
Description: Fetal abdominal circumference by 2-D ultrasound at 35 weeks gestation.
Time Frame: 35 weeks gestation
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Newborn Infants
Number analyzed (Participants) | 47
cm | 32.6 (2.4)

3. Primary Outcome: Estimated Fetal Weight Percentile
Description: Estimated fetal weight percentile by 2-D ultrasound at 35 weeks gestation.
Time Frame: 35 weeks gestation
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Newborn Infants
Number analyzed (Participants) | 47
Percentile | 60.8 (4.7)

ADVERSE EVENTS:
Arm/Group | All Infants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes